CLINICAL TRIAL: NCT05310552
Title: Elucidating Age-related Comorbidity Patterns in Down Syndrome (DS): Prospective Cohort (GO-DS21 Cohort Study)
Brief Title: Elucidating Age-related Comorbidity Patterns in Down Syndrome (DS)
Acronym: GO-DS21
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Fondation Jérôme Lejeune (Other); Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: GODS21CS
Record Dates: First submitted 2022-02-10; First posted 2022-04-05 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Trisomy 21; Obesity; Comorbidities
MeSH Terms: conditions — Down Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples for DNA, RNA on selected participants Plasma and serum samples on those that agreed to donate blood samples Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No interventions - observational study — No interventions - observational study

SUMMARY:
This study is a non-drug, multicenter, prospective cohort study. It will be conducted in 300 volunteers from 12 to 45 years of age (inclusive) with a diagnosis of Down syndrome from 3 countries (France, Spain, United Kingdom (UK)). The basic hypotheses of the study are the following:

1. Diseases (and comorbidity) arise from one or more biological networks perturbed by the genetic disorder (trisomy 21) through interaction with environmental risks factors and epigenetic changes.
2. Health comorbidity patterns in DS individuals (particularly of obesity and related conditions) will likely vary by age and sex.
3. Obesity comorbidity patterns will relate to variation in factors including lifestyle, stress-response, severity of intellectual disability (ID) and variation in cognitive domains such as executive functioning.
4. Stress responses, as measured with cortisol concentrations, will differentiate individuals with DS who are obese and those who are not. Extremes in phenotype (Obese vs. Non-obese) will be related to differences in the metabolomic, transcriptomic, and microbiome concentrations.

DETAILED DESCRIPTION:
The study will be conducted in n= 300 volunteers with DS from 3 countries (France, Spain, UK); equal numbers in 3 age groups (12 - 18 years; 19 - 34 years; 35 - 45 years). The total number of volunteers expected to be included in each country is n = 100.

From the initial cross-sectional cohort, individuals will be selected on the basis of obesity status and invited to participate in a nested case-control study (n = 30 for normal weight DS individuals and n = 30 DS individuals with extreme phenotype). In adults, normal weight is defined as BMI 18.5 to 24.9 and significant obesity as BMI > 35 kg/m2. In children under age 18, the research team will use the International Obesity Task Force (IOTF) curves which are international norms) with IOTF > 30 for obese and IOTF 18.5 - 25 for the normal weight group. The research team will monitor allocation using monthly eCRF recruitment reports for central allocation of recruits to ensure balance between age, sex and BMI between the "cases" and the "controls".

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 12 to 45 years
* With established genetic diagnosis of Down syndrome (full trisomy 21; based on karyotype results - not exclusion if not available but will need to confirm karyotype if not done previously)
* Availability of parent/caregiver to accompany the subject to clinical visits and to be willing to give written informed consent, when necessary

Exclusion Criteria:

* Confirmed mosaic trisomy 21, partial trisomy 21, or translocation
* Comorbid conditions - Participation is allowed as long as the condition(s) are considered stable and it do not interfere with the participation of the study
* Subjects with evidence of dementia or meeting clinical diagnoses for dementia
* Participation in a medication treatment trial in the last 3 months prior to the study

Ages: 12 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: A sample of 300 individuals aged 12-45 years with a diagnosis of Down syndrome will be recruited within the 3 sites.
  Participants will be recruited in three age groups stratified by sex:
  * Adolescents (12-18 years; n = 100)
  * Young adults (19-34 years; n = 100)
  * Middle-age adults (35-45 years; n = 100).
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 1 year
  Height and weight measurements will be aggregated to arrive at one reported value: Body Mass Index (BMI), in kg/m^2
Food Frequency Questionnaire | 1 year
  Average daily nutrient intake
Short Minnesota Leisure Time Physical Activity Questionnaire | 1 year
  Energy expenditure in 14 days
Mental health questionnaire | 1 year
  Reiss Screen for Maladaptive Behaviour - composite outcome measure consisting of the following multiple sub-measures:
  * Aggressive behavior
  * Autism
  * Psychosis
  * Paranoia
  * Depression (behavioural signs)
  * Depression (physical signs)
  * Dependent personality disorder
  * Avoidant disorder

CONTACTS AND LOCATIONS:
Locations (3):
- Institute Jérôme Lejeune, Paris, France
- Institut Hospital del Mar d'Investigacions Mèdiques, Barcelona, Spain
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will be shared within the GO-DS21 Consortium.

REFERENCES:
- See also: GO-DS21 Consortium webpage — https://go-ds21.eu/project/our-vision/